CLINICAL TRIAL: NCT06545396
Title: Characterization Of The Efficacy And Safety Of Illumination Dose Reduction In Red Light Photodynamic Therapy For The Treatment Of Actinic Keratoses And Their Cancerization Field
Brief Title: Efficacy And Safety Of Illumination Dose Reduction In Red Light Photodynamic Therapy For Actinic Keratoses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Jorge Naharro-Rodriguez, Principal Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 154/23
Record Dates: First submitted 2024-08-03; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Actinic Keratoses
Keywords: Photodynamic therapy
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional photodynamic therapy with red light and methyl aminolevulinate (Active Comparator): PDT exposing the area to a red light source for 8 minutes with a spectrum of 630 nm and 37J/cm2, with the illumination intensity being less than 200 mW/cm2.
  Interventions: Other: Full-dose illumination protocol
- Half-dose illumination protocol photodynamic therapy with red light and methyl aminolevulinate (Experimental): PDT exposing the area to a red light source for 8 minutes with a spectrum of 630 nm and 18,5J/cm2, with the illumination intensity being less than 200 mW/cm2.
  Interventions: Other: Half-dose illumination protocol

INTERVENTIONS:
Other: Half-dose illumination protocol — Area will be treated according to the classic protocol, in a single session. First, the surface of the actinic keratoses will be scraped to remove scales and crusts. Using a spatula, a sufficient amount of photosensitizing cream will be applied to cover the treatment area (1 mm thick). The treated area will then be covered with an occlusive dressing for 3 hours. After this interval, the dressing will be removed and the area will be exposed to a red light source for 8 minutes with a spectrum of 630 nm and 18,5J/cm2, with the illumination intensity being less than 200 mW/cm2.
  Arms: Half-dose illumination protocol photodynamic therapy with red light and methyl aminolevulinate
Other: Full-dose illumination protocol — Area will be treated according to the classic protocol, in a single session. First, the surface of the actinic keratoses will be scraped to remove scales and crusts. Using a spatula, a sufficient amount of photosensitizing cream will be applied to cover the treatment area (1 mm thick). The treated area will then be covered with an occlusive dressing for 3 hours. After this interval, the dressing will be removed and the area will be exposed to a red light source for 8 minutes with a spectrum of 630 nm and 37J/cm2, with the illumination intensity being less than 200 mW/cm2.
  Arms: Conventional photodynamic therapy with red light and methyl aminolevulinate

SUMMARY:
The goal of this clinical trial is to compare the tolerance and efficacy of conventional photodynamic therapy (PDT) with red light versus PDT with red light at half dose of illumination, as well as the changes produced by both interventions at the biomolecular level in patients with multiple actinic keratosis on the scalp. The main questions it aims to answer are:

Does PDT with half-dose illumination protocol maintain clinical and biomolecular efficacy?

Does PDT with half-dose illumination protocol improve intervention tolerance?

Researchers will compare both treatment protocols using the patient as its own control.

Participants scalp will be divided in two halves, one will be treated with PDT at conventional doses and the other with the half-dose illumination protocol, a skin biopsy will be obtained both pre and post-treatment of each of the areas. Variables will be assessed during the 3 visits of the study.

DETAILED DESCRIPTION:
The goal of the clinical trial is to compare efficacy and tolerance of photodynamic therapy (PDT) with red light at half dose illumination protocol with conventional PDT for the treatment of grade I and II actinic keratosis. The main hypotheses is that half-light protocol PDT could maintain efficacy while improving tolerance of the procedure.

With this aim the investigators will compare the efficacy of the clinical response after field treatment with photodynamic therapy with red light at half dose versus conventional photodynamic therapy with standard red light in patients with scalp actinic keratoses as well as determine changes in molecular biomarkers at the histological and immunohistochemical level pre- and post-treatment with conventional PDT and PDT with red light at half dose.

The included patients will have their scalp divided into two halves of similar size using the interparietal line as a separation method; one half will be treated with conventional PDT and the other half with half-dose PDT. This is a comparative study between two treatment modalities, both of which will be applied to all patients, and in half of the sample, four skin biopsies of the affected area (two pre and tw post-treatment) will also be performed to conduct an immunohistochemical analysis of the skin samples. Both treatment protocols will be compared using the patient as his or her own protocol. Variables will be assessed during the 3 visits of the study (baseline, 3 months and 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patient with grade I and II actinic keratoses (AK) of Olsen on the scalp requiring field cancerization treatment.
* ≥ 18 years old.
* More than 5 AK per field of cancerization to be treated.
* More than 6 months since the last field treatment for AK performed.
* No AK in clinical grade III progression of Olsen or showing signs suggestive of being invasive squamous cell carcinoma.

Exclusion Criteria:

* Patients with photodermatoses.
* Patients sensitive to methyl-aminolevulinate.
* Patients with disabilities or unable to provide informed consent.
* Patients who do not tolerate or do not wish to be treated with PDT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Response of 75% of the treated actinic keratosis at 3 months post-intervention. | 3 months after de procedure
  Total count of actinic keratosis will be assessed

SECONDARY OUTCOMES:
Tolerance during intervention | During the procedure
  Pain assessed by Visual Analogue Scale (VAS), from 0 (no pain) to 10 (worst pain)
Histological grade of actinic keratosis in biopsies as well as relevant biomarkers | 3 months after the procedure
  E-cadherin, MMPs, p53, UEA, HSP47 and CD117/c-kit presence on the tissue (from + to +++, depending on the intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Naharro-Rodriguez, M.D., Principal Investigator — No organization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trakatelli M, Ulrich C, del Marmol V, Euvrard S, Stockfleth E, Abeni D. Epidemiology of nonmelanoma skin cancer (NMSC) in Europe: accurate and comparable data are needed for effective public health monitoring and interventions. Br J Dermatol. 2007 May;156 Suppl 3:1-7. doi: 10.1111/j.1365-2133.2007.07861.x. PMID 17488399
- [Result] Rowert-Huber J, Patel MJ, Forschner T, Ulrich C, Eberle J, Kerl H, Sterry W, Stockfleth E. Actinic keratosis is an early in situ squamous cell carcinoma: a proposal for reclassification. Br J Dermatol. 2007 May;156 Suppl 3:8-12. doi: 10.1111/j.1365-2133.2007.07860.x. PMID 17488400
- [Result] Wheller L, Soyer HP. Clinical features of actinic keratoses and early squamous cell carcinoma. Curr Probl Dermatol. 2015;46:58-63. doi: 10.1159/000366536. Epub 2014 Dec 18. PMID 25561207
- [Result] Siegel JA, Korgavkar K, Weinstock MA. Current perspective on actinic keratosis: a review. Br J Dermatol. 2017 Aug;177(2):350-358. doi: 10.1111/bjd.14852. Epub 2016 Aug 8. PMID 27500794
- [Result] Chen SC, Hill ND, Veledar E, Swetter SM, Weinstock MA. Reliability of quantification measures of actinic keratosis. Br J Dermatol. 2013 Dec;169(6):1219-22. doi: 10.1111/bjd.12591. PMID 24033340
- [Result] Schmitz L, Gupta G, Stucker M, Doerler M, Gambichler T, Welzel J, Szeimies RM, Bierhoff E, Stockfleth E, Dirschka T. Evaluation of two histological classifications for actinic keratoses - PRO classification scored highest inter-rater reliability. J Eur Acad Dermatol Venereol. 2019 Jun;33(6):1092-1097. doi: 10.1111/jdv.15580. Epub 2019 Apr 3. PMID 30887613
- [Result] Willenbrink TJ, Ruiz ES, Cornejo CM, Schmults CD, Arron ST, Jambusaria-Pahlajani A. Field cancerization: Definition, epidemiology, risk factors, and outcomes. J Am Acad Dermatol. 2020 Sep;83(3):709-717. doi: 10.1016/j.jaad.2020.03.126. Epub 2020 May 7. PMID 32387665
- [Result] Fernandez-Guarino M, Fonda Pascual P, Lizuain Gomez P, Harto Castano A, Jaen Olasolo P. Split-face study comparing conventional MAL photodynamic therapy in multiple actinic keratosis with complete time vs. half-time red light LED conventional illumination. J Eur Acad Dermatol Venereol. 2019 Aug;33(8):1529-1534. doi: 10.1111/jdv.15566. Epub 2019 Apr 15. PMID 30868672
- [Result] Novak B, Heesen L, Schary N, Lubbert H. The influence of different illumination parameters on protoporphyrin IX induced cell death in squamous cell carcinoma cells. Photodiagnosis Photodyn Ther. 2018 Mar;21:385-392. doi: 10.1016/j.pdpdt.2018.02.007. Epub 2018 Feb 7. PMID 29427796
- [Result] Campione E, Di Prete M, Di Raimondo C, Costanza G, Palumbo V, Garofalo V, Mazzilli S, Franceschini C, Dika E, Bianchi L, Orlandi A. Topical Treatment of Actinic Keratosis and Metalloproteinase Expression: A Clinico-Pathological Retrospective Study. Int J Mol Sci. 2022 Sep 26;23(19):11351. doi: 10.3390/ijms231911351. PMID 36232651
- [Result] Bobyr I, Campanati A, Consales V, Martina E, Molinelli E, Diotallevi F, Brisigotti V, Giangiacomi M, Ganzetti G, Giuliodori K, Offidani A. Ingenol mebutate in actinic keratosis: a clinical, videodermoscopic and immunohistochemical study. J Eur Acad Dermatol Venereol. 2017 Feb;31(2):260-266. doi: 10.1111/jdv.13831. Epub 2016 Jul 25. PMID 27453064